CLINICAL TRIAL: NCT03152994
Title: The Early Predictors,Neutrophil-lymphocyte Ratio (NLR), Platelet-lymphocyte Ratio (PLR) and Lymphocyte-monocyte Ratio (LMR) for Developing Type 2 Diabetes Mellitus in Stable Patients With Chronic Obstructive Pulmonary Disease
Brief Title: The Early Predictors for Developing Type 2 Diabetes Mellitus in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CX0422
Record Dates: First submitted 2017-05-01; First posted 2017-05-15 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2017-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Type 2 Diabetes Mellitus
Keywords: Chronic Obstructive Pulmonary Disease; Type 2 Diabetes Mellitus; neutrophil-lymphocyte ratio; platelet-lymphocyte ratio; lymphocyte-monocyte ratio
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients with T2DM: For it's an observational study, fasting blood glucose(FBG) will be checked every six months. The patients who will develope T2DM during the follow-up will be divided into the group"COPD patients with T2DM".
  Interventions: Other: Checking fasting blood glucose(FBG)
- COPD patients without T2DM: For it's an observational study, fasting blood glucose(FBG) will be checked every six months. The patients who won't develope T2DM during the follow-up will be divided into the group"COPD patients without T2DM".
  Interventions: Other: Checking fasting blood glucose(FBG)

INTERVENTIONS:
Other: Checking fasting blood glucose(FBG) — This is an observational study,fasting blood glucose(FBG) of each patient will be checked every six months.

SUMMARY:
Chronic obstructive pulmonary disease(COPD), characterized by persistent airflow limitation, associated with an progressive chronic inflammatory response of the lung to noxious particles or gases, can lead to dyspnea and limited mobility and influence the life quality of patients severely. Type 2 diabetes mellitus(T2DM), as a common complication of COPD, has got more attention in comprehensive control of COPD. Stress response and metabolic disorder are more likely to happen in COPD patients with T2DM in high level inflammation status, which decrease the drug efficacy, increase the risk of acute exacerbation of COPD, complications and mortality.

Both COPD and T2DM are chronic inflammatory disease with long term, there is close relationship in occurrence and development of each other, and the patients with severe COPD are more likely to develop T2DM. Monitoring the acute inflammation maker of C reactive protein (CRP) and IL-6(interleukin-6) is the most useable way to predict the inflammatory status and condition of COPD patient with T2DM, however the chronic inflammation maker is lacking. Neutrophil-to-Lymphocyte ratio(NLR), platelet-lymphocyte ratio (PLR) and lymphocyte-monocyte ratio (LMR) , the new, cheap and easy-tested chronic inflammatory markers, have got great research in early predicting the tumor such as nasopharyngeal carcinoma, soft tissue sarcoma and small-cell lung cancer,among them, NLR has manifest promising application in predicting insulin-resistance. However the value about NLR,PLR and LMR to predict the T2DM in COPD patients remain unknown and many articles related to NLR and COPD are retrospective.

The investigators attempt to analyze the risk factors and predict value of NLR,PLR and LMR about developing T2DM in COPD patients with prospective method.

DETAILED DESCRIPTION:
All the subjects will experience the follow-up every six months, accompanying the monitoring of fast blood glucose (FBG). The complete follow-up will span three years. The follow-up for one patient will stop early when its FBG≥7.0mmol/L which indicates the patient has developed new T2DM.

The subjects will be divided into two groups according to whether patients develop T2DM at the end of each follow-up, namely, COPD patients with T2DM and COPD patients without T2DM

ELIGIBILITY:
Inclusion Criteria:

* The patients diagnosed with stable COPD but no T2DM between April 2017 to April 2020 at Zhu Jiang Hospital of Southern Medical University, will be included.

The diagnosis of COPD is according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2017 Report.

T2DM diagnosis in accordance with the diagnostic criteria of WHO1999.

Exclusion Criteria:

* Patients will be excluded if they have other chronic or acute respiratory disease except COPD, such as bronchiectasia, lung tumor, interstitial pneumonia and hydrothorax; bilateral pulmonary multiple bullae; with metabolic disease such as T2DM, hyperthyroidism or hypothyroidism; questionnaire and laboratory dada was incomplete; with infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients diagnosed with stable COPD but no T2DM between April 2017 to April 2020 at Zhujiang Hospital of Southern Medical University, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
fasting blood glucose(FBG) | Change from baseline in FBG(month 6, month 12, month 18, month 24, month 30, month 36)
  FBG≥7.0mmol/L indicates the patient have developed new T2DM.

SECONDARY OUTCOMES:
routine blood parameters（composite outcome measure） | For the patients who will develop T2DM during the follow up, to be tested at baseline and the time of outcome 1(FBG)≥7.0 (month 6, month 12, month 18, month 24, month 30 or month 36); For others, at baseline and the end of study(month 36)
  The value of neutrophil-lymphocyte ratio (NLR), platelet-lymphocyte ratio (PLR) and lymphocyte-monocyte ratio (LMR) will be calculated by counting neutrophil, lymphocyte, platelet and monocyte in blood.
inspiratory muscle function（composite outcome measure） | For the patients who will develop T2DM during the follow up, to be tested at baseline and the time of outcome 1(FBG)≥7.0 (month 6, month 12, month 18, month 24, month 30 or month 36); For others, at baseline and the end of study(month 36)
  Currently, a variety of methods can be used to evaluate respiratory muscle function,including maximal inspiratory(PImax),expiratory pressures(PEmax)
blood biochemistry（composite outcome measure） | For the patients who will develop T2DM during the follow up, to be tested at baseline and the time of outcome 1(FBG)≥7.0 (month 6, month 12, month 18, month 24, month 30 or month 36); For others, at baseline and the end of study(month 36)
  including HbA1c, triglycerides(TG), total cholesterol(TC), HDL-C, LDL-C, C-reactive protein(CRP), ESR(erythrocyte sedimentation rate), albumin.
Exercise capacity (composite outcome measure) | For the patients who will develop T2DM during the follow up, to be tested at baseline and the time of outcome 1(FBG)≥7.0 (month 6, month 12, month 18, month 24, month 30 or month 36); For others, at baseline and the end of study(month 36)
  Exercise capacity is evaluated using the 6-min walking distance(6MWD) according to American Thoracic Society guidelines.

OTHER OUTCOMES:
Symptom Evaluation(composite outcome measure) | For the patients who will develop T2DM during the follow up, to be tested at baseline and the time of outcome 1(FBG)≥7.0 (month 6, month 12, month 18, month 24, month 30 or month 36); For others, at baseline and the end of study(month 36)
  Individuals with chronic respiratory disease often have symptoms such as dyspnea, fatigue, cough, weakness and psychological distress. Instruments for assessment of multiple symptoms include COPD Assessment Test(CAT) and Modified Medical British Research Council Scale(mMRC).

CONTACTS AND LOCATIONS:
Overall Officials: Xin Chen, Doctor, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital,Southern Medical Universicity, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided